CLINICAL TRIAL: NCT00096811
Title: A Treatment Use Protocol of Entecavir in Subjects With Chronic Hepatitis B Infection Who Have Failed or Who Are Intolerant of Available Therapies
Brief Title: Entecavir for Subjects With Chronic Hepatitis B Infection: An Early Access Program
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-900
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B; Chronic Disease
MeSH Terms: conditions — Hepatitis B; Chronic Disease | interventions — entecavir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 1 mg once daily. Until subject achieves a complete response or until ETV approved and marketed in a given country.
  Other Names: Baraclude

SUMMARY:
The purpose of this clinical research study is to provide entecavir to subjects with chronic Hepatitis B infection who have failed or who have demonstrated intolerance of marketed therapies or for those in whom use of these agents is contraindicated and that have no other available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis B Early Access Program

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Israel (5):
  - Local Institution, Jerusalem
  - Local Institution, Nazareth
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv